CLINICAL TRIAL: NCT06975137
Title: Adapting an Evidenced-based Intervention to Reduce IPV for Use Among Young Heterosexual Couples in South Africa - Zithandani SSCF - Phase 2: Pilot
Brief Title: Zithandani Stepping Stones and Creating Futures - Phase 2 Pilot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: Medical Research Council, South Africa (Other); University College, London (Other); Project Empower (Other)
Responsible Party: Principal Investigator, Andrew Gibbs, Senior Lecturer, University of Exeter
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1633030; MR/X004090/1 (Other Grant/Funding Number: UKRI)
Record Dates: First submitted 2025-05-07; First posted 2025-05-16 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Intimate Partner Violence (IPV); Earning Outcomes; Mental Health; Couple Communication; Couple Conflict; Couples; Livelihoods
Keywords: informal settlements; South Africa; couples; intimate partner violence; couples communication; mental health; livelihoods
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zithandani Stepping Stones and Creating Futures (Experimental): Couples intervention delivered in groups of 4-7 heterosexual couples.
  Interventions: Behavioral: Zithandani Stepping Stones and Creating Futures

INTERVENTIONS:
Behavioral: Zithandani Stepping Stones and Creating Futures — Delivered to heterosexual couples. 14 group based sessions, with each session lasting approximately 3 hours. Sessions are delivered by two trained facilitators. Intervention focused on transforming gender norms, strengthening communication, reducing symptoms of poor mental health and improving relationship dynamics. Mixture of couples focused, same-gender discussions, and whole group discussions.

SUMMARY:
The goal of this uncontrolled intervention study is to assess whether Zithandani Stepping Stones and Creating Futures is feasible to deliver, acceptable for participants, safe for participants and to estimate effect sizes, in young (ages 18-40 years) heterosexual couples, living in urban informal settlements in eThekwini Municipality, South Africa. The main questions it aims to answer are:

1. Is Zithandani SSCF feasible to deliver to young couples, and what are the barriers and opportunities in intervention delivery?
2. Is Zithandani SSCF acceptable to participants? What do they like and what do they not like about the intervention?
3. Is Zithandani SSCF safe for female participants and do they engage adequately?
4. Does Zithandani SSCF show indication of positive change on key indicators and what are the effect sizes?

Participants will be recruited as heterosexual couples and participate in 14 sessions, each approximately 3 hours long, with between 4 and 6 other couples, focused on gender norms, livelihoods and communication.

ELIGIBILITY:
Individual inclusion:

* Aged 18-40 years,
* Reside in the selected community
* Not in full time permanent employment, or in full-time education
* Able to communicate in the main languages of the study (English, isiXhosa or isiZulu)
* Able and willing to provide informed consent to participate

Joint inclusion criteria:

* Be a heterosexual couple
* Been together in a relationship for a minimum of 6 months
* Relationship is public knowledge
* Willing to participate in an intervention

Exclusion criteria individuals is as follows:

* Under 18 or 41+ years old
* Planning on leaving the community in the next 3 months
* Unable or unwilling to provide informed consent
* Unable to communicate in the main study languages

Joint couples exclusion criteria

* Relationship is not public knowledge
* Have been together for less than 6 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Physical IPV | 6 months post baseline
  Self-reports focused on men's perpetration and women's experience of physical intimate partner violence in the past 3 months, based on the WHO Violence Against Women Module - with 5 items. Recoded as a binary (yes/no)
Sexual IPV | 6 months post baseline
  Self-reports focused on men's perpetration and women's experience of sexual intimate partner violence in the past 3 months, based on the WHO Violence Against Women Module - with 3 items. Recoded as a binary (yes/no)
Emotional IPV | 6 months post baseline
  Self-reports focused on men's perpetration and women's experience of sexual intimate partner violence in the past 3 months, based on the WHO Violence Against Women Module - with 8 items. Recoded as a binary (yes/no)
Economic IPV | 6 months post baseline
  Self-reports focused on men's perpetration and women's experience of sexual intimate partner violence in the past 3 months, based on the WHO Violence Against Women Module - with 7 items. Recoded as a binary (yes/no)

SECONDARY OUTCOMES:
Gender Attitudes | 6 months post baseline
  Attitudes in relation to gender and acceptability of violence (9 items) based on prior research in South Africa. Responses (Strongly Disagree to Strongly Agree) range 9-45, higher scores indicative of greater inequitable gender attitudes.
Violence towards children | 6 months post baseline
  Among those reporting a child living in their home, perpetration of physical and/or emotional abuse in the past 4 weeks against the child, using 4 items. Recoded into yes/no.
Trust in relationship/partner measured using the Dyadic Trust scale | 6 months post baseline
  8 Items forming the Dyadic Trust (Larzelere & Huston, 1980), summed with range 8-45. Higher scores indicate more trust in relationship/partner.
Relationship Satisfaction | 6 months post baseline
  5 items (Woolf-King et al., 2019) focused on satisfaction in relationship, with scores from 0-50, and higher scores indicate greater satisfaction in relationship.
Fear of Emotional Intimacy | 6 months post baseline
  35 items, from (Descutner & Thelen, 1991) responses Strongly Disagree to Strongly Agree (5 point Likert), range 35-175. Higher scores indicate greater fear of emotional intimacy.
Empathy for Partner assessed with the Interpersonal Reactivity Index for Couples (IRIC) scale. | 6 months post baseline
  13 items, Empathetic concern using the Interpersonal Reactivity Index for Couples (IRIC) scale. (Péloquin & Lafontaine, 2010) summed together to create score. Score range: 0-52, with higher scores indicating greater empathy for partner.
Sexual Intimacy | 6 months post baseline
  13 items, drawn from Conroy et al. (2021), developed in Malawi, and previously used in South Africa. Responses: Strongly disagree to strongly agree (4 point Likert response). Individual items summed together to create a continuous score (13-52). Higher scores indicative of greater sexual intimacy
Communication with partner assessed using the Communications Pattern Questionnaire | 6 months post baseline
  11 items, from the Communications Pattern Questionnaire and previously used in South Africa (Woolf-King et al., 2019). Range 11-55, higher scores indicate 'better' communication with partner.
Depressive Symptoms assessed using the Patient Health Questionnaire - 9 (PHQ9) | 6 months post baseline
  Patient Health Questionnaire - 9 (PHQ9) asking about past 2 week symptoms of depression. Range 0-27. Higher scores indicative of more symptoms of depression.
Anxiety Symptoms assessed using the Generalised Anxiety Disorder 7 (GAD7) questionnaire | 6 months post baseline
  Generalised Anxiety Disorder 7 (GAD7) (Spitzer et al., 2006) asking about past 2 weeks symptoms of anxiety. Range 0-21. Highers scores indicative of more symptoms of anxiety.
Emotional Dysregulation assessed using the Difficulties in Emotional Regulation Scale 16 | 6 months post baseline
  Difficulties in Emotional Regulation Scale 16 (DERS-16) - 16 items (Bjureberg et al., 2016) adapted for use in South Africa. Range 16-80, with higher scores indicating greater emotional dysregulation.
Alcohol Consumption in past 3 months, assessed with modified Alcohol use disorders identification test consumption (AUDIT C) | 6 months post baseline
  Alcohol use disorders identification test consumption (AUDIT C) (3 items). Rather than asking about past 12 months as is normal, items reworded to ask about past 3 months (e.g. In the last 3 months, how often do you have a drink containing alcohol?). Response options as in original scale. Scores range from 0-13, with higher scores indicating more alcohol consumption.
Earnings in past month | 6 months post baseline
  A single item question asks "Considering all the money you earned from jobs or selling things (excluding grants), how much did you earn last month?" Responses are in Rands (ZAR) and a continuous scale, with no upper limit.
Money participant saved in past month | 6 months post baseline
  A single item question asks "In the last month how much did you put aside for savings?" Responses are in Rands (ZAR) and are on a continuous scale, with no upper limit.
Hunger in the past month | 6 months post baseline
  Household food-security questionnaire (3 items) asking about hunger in the household in the past 4 weeks. Range 3-12 with higher scores indicative of greater food insecurity.
Frequency of work efforts | 6 months post baseline
  7 items asking about work effort in the past 3 months, adapted for use in South Africa. Scored 0-3, with range 0-21, with higher scores indicative of greater livelihoods effort.

OTHER OUTCOMES:
Individual Attendance at Intervention | From enrollment to end of intervention deliver at ~7 weeks
  Proportion of sessions attended by individuals who provide informed consent.
Couples Attendance at Intervention | From enrollment to end of intervention deliver at ~7 weeks
  Proportion of sessions attended by couples who provide informed consent.

CONTACTS AND LOCATIONS:
Locations (1):
- South African Medical Research Council, Durban, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared at data repository 12 months after data collection is completed. Data will either be at the SAMRC data repository or the UK Data Service.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after study completion.
Access Criteria: Free to download once registered on appropriate sites.